CLINICAL TRIAL: NCT06639152
Title: A Comparative Study on the Effect of Oil-based Versus Water-based Contrast Agents in Hysterosalpingography on Improving the Ongoing Pregnancy Rate in Infertile Women: a Prospective Cohort Study.
Brief Title: Oil-based Vs. Water-based Contrast Medium in Hysterosalpingography for Infertile Women in Improving Fertility Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Peace Maternity and Child Health Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GKLW2018-23
Record Dates: First submitted 2024-09-29; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2018-12

CONDITIONS: Infertility
Keywords: Infertility; Hysterosalpingography; Fertility outcome; oil-based contrast medium; water-based contrast medium
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Participants were divided into those who received an oil-based contrast medium (ethiodized poppyseed oil) and a water-based contrast medium (Ioversol) based on a shared medical decision-making process between patients and healthcare providers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oil-based contrast medium (Experimental): oil-based contrast medium: ethiodized poppyseed oil (Jiangsu Hengrui Medicine Co., Ltd., Lianyungang, Jiangsu Province, China, H20067895, iodine concentration of 480 mg/ml)
  Interventions: Drug: oil-based contrast medium
- warer-based contrast medium (Active Comparator): water-based contrast medium: Ioversol (Jiangsu Hengrui Medicine Co., Ltd., Lianyungang, Jiangsu Province, China, H20067895, iodine concentration of 320 mg/ml)
  Interventions: Drug: water-based contrast medium

INTERVENTIONS:
Drug: oil-based contrast medium — In oil group, ethiodized poppyseed oil (Jiangsu Hengrui Medicine Co., Ltd., Lianyungang, Jiangsu Province, China, H20067895, iodine concentration of 480 mg/ml) was used as the contrast medium for hysterosalpingography.
  Arms: oil-based contrast medium
Drug: water-based contrast medium — In water group, Ioversol (Jiangsu Hengrui Medicine Co., Ltd., Lianyungang, Jiangsu Province, China, H20067895, iodine concentration of 320 mg/ml) was used as the contrast medium for hysterosalpingography.
  Arms: warer-based contrast medium

SUMMARY:
The goal of this clinical trial is to compare the effects of oil-based contrast medium (OBCM) and water-based contrast medium (WBCM) during hysterosalpingography（HSG）on pregnancy outcomes in infertile women. The main question it aims to answer is whether an oil-based contrast medium improves fertility outcomes in infertile women. Participants were divided into those who received an oil-based contrast medium (ethiodized poppyseed oil) and a water-based contrast medium (Ioversol) based on a shared medical decision-making process between patients and healthcare providers. The two contrast agents used in this study are routinely employed in clinical practice and will not affect the participants' health. Participants are required to complete some clinical questionnaires before and after the HSG procedure to provide clinical information. Other than that, there will be no additional costs for participants.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years
2. infertility for at least one year without the use of contraceptives.

Exclusion Criteria:

1. endocrine disorders, including Cushing's syndrome, hypothalamic amenorrhea, adrenal hyperplasia, diabetes, or thyroid dysfunction (except for well-controlled hypothyroidism with a TSH level between 0.3 and 4.0 mIU/L)
2. known allergy to contrast agents, specifically iodine
3. male partner infertility, defined as post-wash sperm motility <3 million/mL or <1 million/mL without sperm washing
4. contraindications for undergoing HSG
5. refusal to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1187 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
live birth | From enrollment to the end of treatment at 6 months
  The primary outcome measure is live birth from pregnancies occurring within 6 months after HSG, defined as a live birth after 24 weeks of gestation, with the last menstrual period starting within six months post-HSG.

SECONDARY OUTCOMES:
clinical pregnancy | From enrollment to the end of treatment at 6 months
  clinical pregnancy within six months post-HSG, indicated by the detection of a gestational sac on ultrasound
ongoing pregnancy | From enrollment to the end of treatment at 6 months
  ongoing pregnancy within six months after HSG, defined as the presence of a fetal heartbeat on ultrasound after 12 weeks of gestation
miscarriage | From enrollment to the end of treatment at 6 months
  Miscarriage was identified by the absence of a fetal heartbeat on ultrasound or loss before 12 weeks of gestation within 6 months after HSG.
ectopic pregnancy | From enrollment to the end of treatment at 6 months
  Ectopic pregnancy was defined as pregnancy where implantation occurs outside the uterine cavity within 6 months after HSG.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Principal Investigator — International Peace Maternity and Child Health Hospital affiliated to Shanghai Jiao Tong University, School of Medicine
Locations (1):
- International Peace Maternity and Child Health Hospital affiliated to Shanghai Jiao Tong University, School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the publication of the results
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years after the publication of results

REFERENCES:
- [Derived] Zhu Q, Lu M, Liang G, Wang Y, Xia W, Yan L, Sun T, Mol BW, Zhang J. Oil-based vs. water-based contrast medium in hysterosalpingography for older, anovulatory, and infertile women with high-risk of tubal disease. Eur J Obstet Gynecol Reprod Biol. 2025 Sep;313:114651. doi: 10.1016/j.ejogrb.2025.114651. Epub 2025 Aug 11. PMID 40816246